CLINICAL TRIAL: NCT02222818
Title: Cardiac Resynchronization Therapy Efficacy Enhancements
Acronym: CRTee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CRTee
Record Dates: First submitted 2014-08-19; First posted 2014-08-21 (Estimated); Results first posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2016-11

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: CAFR first (Other): Subjects randomized to Group A will receive CAFR first, then cross over to CAFRPlus.
  Interventions: Device: Conducted AF Response (CAFR); Device: Conducted AF Response Plus (CAFRPlus)
- Group B: CAFRPlus first (Other): Subjects randomized to Group B will receive CAFRPlus first, then cross over to CAFR.
  Interventions: Device: Conducted AF Response (CAFR); Device: Conducted AF Response Plus (CAFRPlus)

INTERVENTIONS:
Device: Conducted AF Response (CAFR) — The CAFR algorithm is currently available in the Medtronic market-released devices and intended to promote delivery of CRT pacing during conducted AT/AF episodes.
Device: Conducted AF Response Plus (CAFRPlus) — The CAFRPlus algorithm is part of the CRTee feature set. This feature set has a diagnostic element that tracks the loss of effective CRT pacing that is occurring over time, both during normal sinus rhythm (NSR) and during AF. It also has an interventional element (i.e. CAFRPlus) that uses this evaluation of effective CRT pacing to adjust the pacing rate during AF to decrease loss of effective CRT pacing.

SUMMARY:
The purpose of this study is to demonstrate that the amount of effective CRT (Cardiac Resynchronization Therapy) pacing during AF (atrial fibrillation) when CAFRPlus (Conducted AF Response Plus) is applied is not inferior to the amount of effective CRT pacing during AF when CAFR (Conducted AF Response) is applied.

DETAILED DESCRIPTION:
The CRTee study is an IDE, prospective, multi-center, randomized, controlled, crossover clinical study, conducted worldwide and designed to demonstrate that the amount of effective CRT pacing during AF (atrial fibrillation) when CAFRPlus (Conducted AF Response Plus) is applied is not inferior to the amount of effective CRT pacing during AF when CAFR (Conducted AF Response) is applied.

The study will be conducted at up to 30 centers located in the United States, Europe and Middle East and Africa (MEA).

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing to sign and date the study patient Informed Consent form.
* Subject is at least 18 years of age (or older, if required by local law).
* Subject is expected to remain available after enrollment to complete follow-up visits in both arms of the study
* Subject has had a Medtronic Viva or Brava CRT-D device implanted at least 30 days prior to enrollment.
* Subject has history of AF burden, of at least 6 days of at least 4 hours of AF over any 4 week period within the last 90 days as documented in device diagnostic data OR if subject has no atrial lead (therefore no device diagnostic data) but clinical evidence of high AF burden.
* Subject has demonstrated history of being able to complete Left Ventricular Capture Management (LVCM) documented in device data.
* Subject has a documented % V pacing during AF of less than or equal to 97% within 90 days prior to enrollment or within 10 days after enrollment.

Exclusion Criteria:

* Subject has undergone AV node ablation for treatment of AF.
* Subject has complete or 3rd degree AV block.
* Subject has had an MI within 30 days.
* Subject has medical conditions that limit study participation (per physician discretion).
* Subject is enrolled in one or more concurrent studies that could confound the study results as determined by Medtronic.
* Subject has a limited life expectancy for non-cardiac causes that would not allow completion of the study.
* Subject is pregnant (in the US, all women of child-bearing potential must undergo a pregnancy test within seven days prior to CRTee download).
* Subject meets the exclusion criteria required by local law.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2014-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suneet Mittal, MD, Principal Investigator — Valley Health System
Locations (19):
- United States (10):
  - Cardiac Arrythmia Services, Boca Raton, Florida
  - Iowa Heart Center, West Des Moines, Iowa
  - North Memorial Heart and Vascular, Minneapolis, Minnesota
  - CentraCare, Saint Cloud, Minnesota
  - North Carolina Heart and Vascular, Raleigh, North Carolina
  - Mount Carmel, Columbus, Ohio
  - Oklahoma Heart, Oklahoma City, Oklahoma
  - Berks Cardiology, Reading, Pennsylvania
  - Texas Cardiac Arrhythmia Services, Austin, Texas
  - Kootenai Heart Clinics, Spokane, Washington
- Magyar Honvédség Honvédkorház, Budapest, Hungary
- Italy (3):
  - Policlinico Universitario Agostino Gemelli, Roma
  - Azienda Ospedaliera Bolognini Seriate - Ospedale Bolognini, Seriate
  - Azienda Ospedaliera Cardinale Panico, Tricase
- Prince Sultan Cardiac Center, Riyadh, Saudi Arabia
- Vychodoslovensky ustav srdcovych a cievnych chorob, a.s., Košice, Slovakia
- Mediclinic Panorama, Cape Town, South Africa
- United Kingdom (2):
  - Liverpool Heart and Chest Hospital NHS Foundation Trust, Liverpool
  - he Newcastle upon Tyne Hospitals NHS Foundation Trust - Freeman Hospital, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Plummer CJ, Frank CM, Bari Z, Al Hebaishi YS, Klepfer RN, Stadler RW, Ghosh S, Liu S, Mittal S. A novel algorithm increases the delivery of effective cardiac resynchronization therapy during atrial fibrillation: The CRTee randomized crossover trial. Heart Rhythm. 2018 Mar;15(3):369-375. doi: 10.1016/j.hrthm.2017.10.026. Epub 2017 Nov 11. PMID 29132930

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 71 subjects were enrolled from 22 investigational centers in the United States, Europe and Middle East. The first subject was enrolled on 07 Oct 2014, and last enrollment was on 08 Jan 2016.
Pre-assignment Details: Of the 71 enrolled subjects, 5 did not meet eligibility criteria (AV node ablation - 2, complete heart block - 3) and were exited from the study prior to randomization assignment.
Period: Period 1
Arm/Group | Group A: CAFR First | Group B: CAFRPlus First
Started | 33 (Start of CAFR evaluation period) | 33 (Start of CAFRPlus evaluation period)
Completed | 33 (End of CAFR evaluation period) | 30 (End of CAFRPlus evaluation period)
Not Completed | 0 | 3
Not completed — Eligibility criteria not met | 0 | 3
Period: Period 2
Arm/Group | Group A: CAFR First | Group B: CAFRPlus First
Started | 33 (Start of CAFRPlus evaluation period) | 30 (Start of CAFR evaluation period)
Completed | 33 (End of CAFRPlus evaluation period) | 30 (End of CAFR evaluation period)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects randomized to either Group A (CAFR first) or Group B (CAFRPlus first).
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: CAFR First | Group B: CAFRPlus First | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.7 (11.6) | 72.4 (9.1) | 71.6 (10.4)
Gender [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 29 | 32 | 61
Region of Enrollment [Number; unit: participants]
  Saudi Arabia | 5 | 4 | 9
  Hungary | 4 | 4 | 8
  United States | 14 | 17 | 31
  Italy | 5 | 4 | 9
  United Kingdom | 3 | 3 | 6
  Slovakia | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Effective CRT Pacing During AF (Non-inferiority Test)
Description: The primary objective is to demonstrate that the percent effective CRT pacing during AF when CAFRPlus is applied is not inferior to when CAFR is applied (non-inferiority test).
Time Frame: Up to 4 months
Population: Randomized subjects who had paired measurements available from both CAFR period and CAFRPlus period.
Measure: Mean (Standard Deviation); unit: percentage of effective CRT pacing
Groups:
- CAFR ON: Percentage of effective CRT pacing during AF when CAFR is ON
- CAFRPlus ON: Percentage of effective CRT pacing during AF when CAFRPlus is ON
Arm/Group | CAFR ON | CAFRPlus ON
Number analyzed (Participants) | 54 | 54
percentage of effective CRT pacing | 80.8 (14.3) | 87.8 (7.8)
Statistical Analysis 1: Comparison: CAFR ON vs CAFRPlus ON; Null Hypothesis (Ho): μd ≤ -2% Alternative Hypothesis (Ha): μd > -2% where μd is the paired difference in percent effective CRT pacing during AF between when CAFRPlus is applied and when CAFR is applied, based on subjects' paired measurements from the two cross-over follow-up periods, and -2% is the non-inferiority margin selected based upon clinical judgment; Test type: Non-Inferiority or Equivalence — In order to demonstrate that CAFRPlus is no less effective than CAFR by a non-inferiority margin of 2%, assuming a true paired difference of 6% and a standard deviation of 15% for the paired differences, a sample size of 39 subjects with paired data is required to achieve 90% statistical power using the one-sample t-test for non-inferiority, while controlling the one-sided type I error rate at 0.025; p < 0.0001, t-test, 1 sided — The threshold for statistical significance was 0.0207, determined by the pre-specified alpha spending function accounting for one interim analysis; Mean Difference (Net) = 7.0, 95.86% CI 2-sided [4.5 to 9.5], Standard Deviation 8.7

2. Secondary Outcome: Percentage of Effective CRT Pacing During AF (Superiority Test)
Description: The secondary objective is to demonstrate that the percent effective CRT pacing during AF when CAFRPlus is applied is greater than when CAFR is applied (superiority test).
Time Frame: Up to 4 months
Population: Randomized subjects who had paired measurements available from both CAFR period and CAFRPlus period.
Measure: Mean (Standard Deviation); unit: percentage of effective CRT pacing
Arm/Group | CAFR ON | CAFRPlus ON
Number analyzed (Participants) | 54 | 54
percentage of effective CRT pacing | 80.8 (14.3) | 87.8 (7.8)
Statistical Analysis 1: Comparison: CAFR ON vs CAFRPlus ON; Null Hypothesis (Ho): μd ≤ 0% Alternative Hypothesis (Ha): μd > 0% where μd is the paired difference in percent effective CRT pacing during AF between when CAFRPlus is applied and when CAFR is applied, based on subjects' paired measurements from the two cross-over follow-up periods; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 7.0, 95.86% CI 2-sided [4.5 to 9.5], Standard Deviation 8.7

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout entire study follow-up (from enrollment to study exit). Subjects' follow-up duration ranged from 0 to 5.4 months, with an average of 2.7 ± 1.6 months for all enrolled subjects.
Groups:
- All Enrolled Subjects: All subjects enrolled in the CRTee study.
Arm/Group | All Enrolled Subjects
Serious Adverse Events (participants affected / at risk) | 7/71
Other Adverse Events (participants affected / at risk) | 5/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Subjects (N=71)
Cardiac failure (Cardiac disorders) | 2 (3)
Ventricular arrhythmia (Cardiac disorders) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Subjects (N=71)
Cardiac failure (Cardiac disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, contracts allow investigators to publish study results per the protocol and publication plan. Investigators and Participating Institutions will provide any publication of Study Data generated by PI and/or Participating Institution to Medtronic for review prior to submission to determine if confidential information ("CI") is included and to check for technical correctness. Medtronic may not censor/interfere with the publication beyond the extent necessary to protect CI.